CLINICAL TRIAL: NCT04796571
Title: Care Coordination and Proactive Care to Improve Utilization of Resources and Reduce Expenditure in High Risk Inflammatory Bowel Disease (IBD) Patients
Acronym: CAPTURE IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Twine Clinical Consulting LLC (Unknown)
Responsible Party: Principal Investigator, Peter Higgins, Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HUM00147500
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding of participants was not possible because telephone visits were only offered to participants in the intervention arm. Investigators were blinded to the randomization order, but patients, staff, and providers were not blinded to arm assignment. The investigators who validated the data and performed the data analysis remained blinded to patient group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Care Coordination Arm (Experimental): Patients were assigned an IBD-focused care coordinator who facilitated a symptom-based monitoring algorithm and supported patient navigation to complement usual care.
  Interventions: Behavioral: Proactive Symptom Monitoring and Care Coordination
- Usual Care (No Intervention): Participants in the usual care arm underwent symptom monitoring through regular push notifications to participants to complete a validated PRO instrument through the Epic EMR patient portal or telephone. These notifications were scheduled on a monthly basis. Results of the monthly PRO instrument were available to their treating IBD doctor with interventions at their discretion.
- passive control arn (No Intervention): To explore whether our usual care arm was influenced by the monthly PRO measurements required for examination of our primary outcome, we compared IBD charges, total charges, ED visits, hospitalizations, and medication utilization at 12 months in the usual care arm to a passive control arm consisting of patients who met eligibility criteria, but were not enrolled in the intervention or usual care arms.

INTERVENTIONS:
Behavioral: Proactive Symptom Monitoring and Care Coordination — Patients randomized to the intervention arm were assigned an IBD-focused care coordinator who facilitated a symptom-based monitoring algorithm and supported patient navigation to complement usual care. Symptom monitoring was facilitated through regular push notifications to participants to complete a validated PRO instrument through the Epic EMR patient portal or telephone. These notifications were scheduled on a monthly basis. The IBD-focused care coordinator made two attempts to reach each participant using portal messaging, followed by a phone call to reduce non-response. PRO questionnaires were reviewed by the care coordinator and out of range scores triggered algorithm-based recommendations to the IBD specialist including stricter monitoring of disease activity, behavioral and medication adherence counseling, facilitation of expedited follow-up with treating providers, and referrals to social work, mental health, and gastroenterology-specific behavioral health services.
  Arms: Care Coordination Arm

SUMMARY:
The study team performed a randomized controlled trial to evaluate the efficacy of a care coordination intervention composed of proactive symptom monitoring and algorithm-based triggers to improve patient reported outcomes (PROs) and healthcare expenditures for high-risk patients with IBD. Enrolled patients with IBD were randomized to proactive symptom monitoring with the support of a care coordinator or usual care.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of IBD (with at least 3 office visits)
* followed in GI clinic within 1 year of enrollment
* in top 20th percentile of predicted risk for subsequent healthcare utilization (previously validated model)

Exclusion Criteria:

* non-IBD driver for high utilization (e.g., active cancer undergoing treatment
* A life expectancy of less than one year, were excluded from participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change in patient reported outcome (PRO) scores | 9 months
  Patient Reported Outcome (PRO) measurements were administered on a monthly basis. The validated Crohn's (CD)-PRO or ulcerative colitis (UC)-PRO were used according to the patient's IBD type (Crohn's or ulcerative colitis).
  Both the CD-PRO and UC-PRO are a set of standardized and validated instruments based on the Crohn's Disease Activity Index and Mayo Clinic Score respectively, which includes six domains: daily bowel movements, functional symptoms, systemic symptoms, daily coping, weekly life impact, and weekly emotional impact. Scores are calculated a composite score across all domains where a score of 0 represents no symptom activity and a score of 40 represents the highest possible symptom burden.
  These were not two separate outcomes, rather two independent measurement instruments (scored on the same scale) specific to the patient's IBD-type to address the specific needs/concerns of the patients based on disease type.
IBD-related charges per person | 12 months
  extracted charges where IBD was the primary diagnosis over study period
Total healthcare charges per person | 12 months
  all extracted charges over study period

SECONDARY OUTCOMES:
Emergency Department (ED) visits per person | 12 months
  extracted number of persons experiencing an ED visit over the study period
Proportion of hospitalizations per person | 12 months
  extracted number of persons experiencing hospitalization over the study period
Change in IBD medication utilization | 12 months
  Use of any of the following medications: biologic therapy, immunosuppressant therapy, corticosteroids, narcotics over study period

CONTACTS AND LOCATIONS:
Overall Officials: Peter Higgins, MD, PhD, MSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share this PHI data with the public, however it there is a request, de-identified data could be arranged.

REFERENCES:
- [Derived] Berinstein JA, Cohen-Mekelburg SA, Greenberg GM, Wray D, Berry SK, Saini SD, Fendrick AM, Adams MA, Waljee AK, Higgins PDR. A Care Coordination Intervention Improves Symptoms But Not Charges in High-Risk Patients With Inflammatory Bowel Disease. Clin Gastroenterol Hepatol. 2022 May;20(5):1029-1038.e9. doi: 10.1016/j.cgh.2021.08.034. Epub 2021 Aug 28. PMID 34461298